CLINICAL TRIAL: NCT03586284
Title: Systemic and Topical Antivirals for Control of Cytomegalovirus Anterior Uveitis: Treatment
Brief Title: Systemic and Topical Antivirals for Control of Cytomegalovirus Anterior Uveitis: Treatment Outcomes
Acronym: STACCATO
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding discontinued.
Sponsor: University of California, San Francisco (Other)
Collaborators: Huang Pacific Foundation (Unknown); Khon Kaen University (Other); King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-24396; NCT03576898 (obsolete NCT alias)
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Cytomegalovirus Anterior Uveitis
Keywords: Cytomegalovirus uveitis; Cytomegalovirus endotheliitis; Cytomegalovirus keratouveitis; Cytomegalovirus iridocyclitis
MeSH Terms: interventions — Valganciclovir; Ganciclovir

STUDY DESIGN:
Intervention Model Description: Multicenter, double-masked, randomized, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Oral Valganciclovir (Active Comparator): Oral Valganciclovir 900mg PO BID Topical placebo solution, 1 drop applied 6 times daily
  Interventions: Drug: Valganciclovir Hydrochloride; Drug: Topical placebo
- Topical Ganciclovir 2% (Active Comparator): Topical Ganciclovir 2% solution, 1 drop applied 6 times daily Placebo pills PO BID
  Interventions: Drug: Ganciclovir Sodium; Drug: Placebo Oral Tablet
- Placebo (Placebo Comparator): Topical placebo solution, 1 drop applied 6 times daily Placebo pills PO BID
  Interventions: Drug: Placebo Oral Tablet; Drug: Topical placebo

INTERVENTIONS:
Drug: Valganciclovir Hydrochloride — 21 to 28 days of oral valganciclovir treatment
  Arms: Oral Valganciclovir
Drug: Ganciclovir Sodium — 21 to 28 days of topical ganciclovir solution treatment
  Arms: Topical Ganciclovir 2%
Drug: Placebo Oral Tablet — 21 to 28 days of placebo pill treatment
  Arms: Placebo; Topical Ganciclovir 2%
Drug: Topical placebo — 21 to 28 days of topical placebo treatment
  Arms: Oral Valganciclovir; Placebo

SUMMARY:
Cytomegalovirus (CMV) is generally a latent and asymptomatic infection in healthy, immunocompetent individuals. In immunocompromised patients CMV is well known to cause a retinitis that can lead to blindness. In immunocompetent patients, however, CMV can cause recurrent inflammation in the front of the eye (anterior uveitis). CMV anterior uveitis produces complications including pain, glaucoma, corneal failure, and vision loss. CMV anterior uveitis is commonly misdiagnosed as a non-infectious anterior uveitis and treated as such, which can beget further complications. Diagnosis requires directed polymerase chain reaction (PCR) testing. While antiviral therapy exists for CMV, identifying the appropriate therapy has been challenging because no randomized trials comparing routes of therapy (particularly oral or topical) have been performed. Oral antiviral therapy of CMV carries blood and kidney side effects that requires laboratory monitoring. Topical therapy has been reported to be effective, but no consensus as to the appropriate drug concentration exists.

Here we propose a double-masked randomized controlled clinical trial comparing the efficacy of oral valganciclovir, topical ganciclovir 2%, and placebo for the treatment of PCR-proven CMV anterior uveitis. This pilot study will provide valuable information concerning the treatment of CMV anterior uveitis with oral and topical medications, including effective concentrations and side-effect profile. The information obtained from this study will help inform future larger clinical trials in CMV anterior uveitis.

DETAILED DESCRIPTION:
Recurrent anterior uveitis in immunocompetent individuals can be caused by multiple members of the herpes virus group, including cytomegalovirus (CMV). Repeated bouts of CMV intraocular inflammation can be associated with ocular hypertension, glaucoma, pain, vision reduction or blindness. CMV anterior uveitis is commonly misdiagnosed as a non-infectious anterior uveitis and treated as such, which can beget further complications. Diagnosis requires directed polymerase chain reaction (PCR) testing. While antiviral therapy exists for CMV, identifying the appropriate therapy has been challenging because no randomized trials comparing routes of therapy (particularly oral or topical) have been performed. Currently, CMV anterior uveitis is typically treated with oral valganciclovir in the United States but carries the risk of serious systemic side effects that necessitate laboratory monitoring. There is evidence that suggests topical ganciclovir can be used to treat and prevent recurrences of CMV anterior uveitis, though the appropriate concentration is not well defined. Topical ganciclovir is attractive because it does not require laboratory monitoring, though a unique side effect profile that includes corneal epitheliopathy and conjunctivitis may preclude long-term use. While anterior chamber paracentesis with polymerase chain reaction (PCR) testing demonstrates CMV during an initial flare of inflammation, it is unknown whether repeated recurrences of inflammation are mediated by viral re-infection and replication in the anterior chamber or if a sterile immune response is at play. Consequently, patients may be submitted to many years of oral or topical antiviral therapy. This strategy poses challenges without proper evaluation of the multiple treatment and long-term management approaches. Further studies are needed to elucidate the most appropriate antiviral therapies that balance efficacy and toxicity while treating CMV anterior uveitis.

There are no studies comparing antivirals for the treatment of CMV anterior uveitis. However, multiple studies have utilized PCR to obtain an initial viral load before treating CMV anterior uveitis. The collective initial CMV viral load from these prior studies (39 patients in total) was approximately 600,000 IU/ml. There was minimal variation within studies in terms of initial viral load, but large variation between studies. To control for variability that can arise from different assays used or assays performed at different centers, we will perform all quantitative PCR at the same United States location. Even fewer studies have documented post-treatment viral loads. Many of the post-treatment PCR values showed undetectable viral loads, making it difficult to estimate viral load reduction trends between treatment groups. Of note, the limited data demonstrated that both intravenous ganciclovir and topical ganciclovir 2% groups showed significant and rapid reductions in viral load, almost always resulting in undetectable levels by 12 weeks, and occasionally as rapidly as 2-3 weeks. We identified three patients from the literature with CMV anterior uveitis that had detectable PCR values during the course of treatment. These patients had a 95% average reduction in viral load 14 days after treatment.

We are proposing a double-masked randomized controlled clinical trial comparing the efficacy of oral valganciclovir, topical ganciclovir 2%, and placebo for the treatment of PCR-proven CMV anterior uveitis. The primary outcome will be percent reduction in viral load. We hypothesize that the oral valganciclovir arm will experience the greatest reduction in viral load. Secondary outcomes will include time to clinical quiescence and the effect of pre-enrollment topical corticosteroid use on initial viral load.

This pilot study will provide valuable information concerning the treatment of CMV anterior uveitis with oral and topical medications, including effective concentrations and side-effect profile. The information obtained from this study will help inform future larger clinical trials in CMV anterior uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical impression consistent with CMV anterior uveitis
* Directed PCR positive for CMV OR previous PCR-proven CMV anterior uveitis
* Willingness to use an acceptable method of contraception during the study period (i.e.

pharmacologic, devices, barrier methods) or abstinence.

Exclusion Criteria:

* Patients <18 years of age
* Intermediate or posterior inflammation (involvement of vitreous, choroid, or retina)
* Received antiviral therapy <14 days prior to enrollment
* Received periocular or intraocular corticosteroid injection < 8 weeks prior to enrollment
* Currently taking oral corticosteroids
* Immunocompromised (primary or secondary immunosuppressive disorders)
* Prior immunosuppressive therapy in the past 6 months
* Directed PCR negative for CMV
* Directed PCR positive for herpes simplex virus (HSV) or varicella zoster virus (VZV)
* Planning to conceive during the study period, pregnant or breast-feeding (blood or urine pregnancy test for all females of child-bearing age is mandatory within 4 weeks prior to enrollment)
* Complete blood count with white blood cell, absolute neutrophil, or platelet count lower than the lower limit of reference laboratory normal
* BUN or Cr above the upper limit of reference laboratory normal
* Recent ocular surgery within the past 30 days, or planned surgery within the next 45 days
* Systemic autoimmune disease or ocular condition (besides anterior uveitis) anticipated to dictate or alter treatment course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Gonzales, MD, Principal Investigator — UCSF Proctor Foundation
Locations (4):
- Proctor Foundation, UCSF, San Francisco, California, United States
- Thailand (3):
  - Chulalongkorn University, Bangkok
  - Chiang Mai University, Chiang Mai
  - Khon Kaen University, Khon Kaen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Takhar JS, Joye AS, Somkijrungroj T, Laovirojjanakul W, Lin CP, Lietman TM, Porco TC, Keenan JD, Gebreegziabher EA, Seitzman GD, Rose-Nussbaumer J, Doan TA, Acharya NR, Gonzales JA. A double masked randomised 4-week, placebo-controlled study in the USA, Thailand and Taiwan to compare the efficacy of oral valganciclovir and topical 2% ganciclovir in the treatment of cytomegalovirus anterior uveitis: study protocol. BMJ Open. 2019 Dec 19;9(12):e033175. doi: 10.1136/bmjopen-2019-033175. PMID 31862739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective recruitment at three uveitis centers (UCSF, Chulalongkorn, Khon Kaen) Jan 2020-Mar 2024 during routine care of adults with active anterior uveitis. Eligibility: ≥1+ AC cells and CMV+ by AC PCR; key exclusions: recent antivirals/steroids, systemic IS, HSV/VZV. 51 randomized (1:1:1; site-stratified blocks) to valganciclovir, 2% ganciclovir, or placebo; 47 completed day-7 sampling. Enrollment ended early due to COVID-related delays/funding.
Pre-assignment Details: Adults with active anterior uveitis gave consent, had slit-lamp exam and anterior chamber paracentesis. Local PCR confirmed CMV and excluded HSV/VZV. While awaiting results, candidates received standard-of-care topical steroids/IOP meds. Washouts: no antivirals ≤14 days; no peri/intraocular steroid ≤8 weeks. Eligible participants completed baseline measures, then were randomized via site-stratified, concealed allocation with masked tablets/drops.
Groups:
- Oral Valganciclovir: Oral valganciclovir 900 mg PO BID
- Topical Ganciclovir 2%: Topical ganciclovir 2% 1 drop applied 6 times daily
- Placebo: Topical placebo solution 1 drop applied 6 times daily
Period: Overall Study
Arm/Group | Oral Valganciclovir | Topical Ganciclovir 2% | Placebo
Started | 19 | 15 | 17
Completed | 19 | 13 | 15
Not Completed | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Valganciclovir | Topical Ganciclovir 2% | Placebo | Total
Number analyzed (Participants) | 19 | 15 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (15.2) | 59.3 (9.9) | 51.7 (18.5) | 54.7 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 7 | 24
  Male | 10 | 7 | 10 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 18 | 14 | 16 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in CMV Viral Load
Description: Pre-treatment minus day-7 CMV DNA load in aqueous humor, reported as log10 IU/mL (WHO-standardized qPCR). Positive values indicate reduction.
Time Frame: 7 days
Population: Includes randomized participants with paired baseline and day-7 aqueous qPCR results (oral 19/19, topical 13/13, placebo 15/15).
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Oral Valganciclovir | Topical Ganciclovir 2% | Placebo
Number analyzed (Participants) | 19 | 13 | 15
log10 IU/mL | 0.59 (0.87) | 0.23 (0.59) | 0.04 (0.44)

2. Secondary Outcome: Number of Participants That Achieved Clinical Quiescence
Description: Comparison between arms of percent that achieved clinical quiescence by final visit (anterior chamber cell ≤ 0.5+).
Time Frame: Day 0 to Day 21 (final visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Valganciclovir | Topical Ganciclovir 2% | Placebo
Number analyzed (Participants) | 19 | 13 | 15
Participants | 19 | 13 | 15

3. Secondary Outcome: Effect of Topical Corticosteroid
Description: What effect did topical corticosteroid use prior to enrollment have on pre-treatment viral load (Day 0)
Time Frame: Day 0 (pre-treatment) viral load (IU/mL)
Measure: Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Oral Valganciclovir | Topical Ganciclovir 2% | Placebo
Number analyzed (Participants) | 19 | 13 | 15
IU/mL | 0.10 [-0.06 to 0.26] | 0.10 [-0.06 to 0.26] | 0.10 [-0.06 to 0.26]

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Oral Valganciclovir | Topical Ganciclovir 2% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15 | 0/13

LIMITATIONS AND CAVEATS:
Small sample and early stopping limited power. Baseline imbalances (e.g., prostaglandin use, viral load) required multivariable adjustment. The 7-day endpoint assesses early antiviral activity and does not address durability, recurrence, or long-term IOP control. Variable aqueous volume made low-end quantitation imprecise; values below the assay's LLOQ were treated as non-quantifiable and set to the LLOQ for analysis. Inference emphasizes adjusted between-arm contrasts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT03586284/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT03586284/SAP_001.pdf